CLINICAL TRIAL: NCT00277225
Title: A Phase I,Randomized, Double Blind, Placebo Controlled Study to Assess the Pharmacokinetics, Immunogenicity and Safety of Escalating Doses of BMS-188667 Given as a Single Intravenous Infusion to Patients With Psoriasis Vulgaris
Brief Title: A Study to Assess the Pharmacokinetics, Immunogenicity and Safety of Escalating Doses of BMS-188667 Given as a Single Intravenous Infusion to Patients With Psoriasis Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-003
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Abatacept

INTERVENTIONS:
Drug: Abatacept

SUMMARY:
The purpose of this protocol is to determine the single-dose pharmacokinetics and immunogicity of BMS-188667 administered as a 1 hour intravenous infusion with extended pharmacokinetic sampling. Safety of all subjects will be assessed in a double blind fashion through the inclusion of placebo controls at each dose level.

ELIGIBILITY:
Inclusion Criteria:

* Subjects required to have a know diagnosis of psoriasis vulgaris involving 5-49% of total body surface area (BSA) for at least six months prior to randomization.
* Subjects clinically insignificant abnormal laboratory or ECG test results who were otherwise healthy and met all remaining eligibility criteria.

Exclusion Criteria:

* Evidence of active bacterial or viral infections at the time of enrollment, including any history of or clinical evidence of infection with Human Immunodeficiency virus (HIV) Hepatitis B or Hepatitis C.
* Any underlying metabolic, hematologic, pulmonary, cardiac, renal hepatic, infectious, psychiatric or gastrointestional condition, which in the opinion of the investigator, placed the subject at unacceptable risk from participation in a study with potentially immunosuppresive therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 1995-11; Primary Completion 1996-06 (Actual); Study Completion 1996-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics throughout study period | Until Day 43 or Day 120 depending on dose level

SECONDARY OUTCOMES:
Safety and Immunogenicity throughout study period. | Until Day 43 or Day 120 depending on dose level and duration of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ralph D. Beasom, M.D., Study Chair — California Institutional Review Board
Locations (1):
- California Clinical Trials Medical Group, Beverly Hills, California, United States